CLINICAL TRIAL: NCT06982625
Title: Supra Inguinal Fascia Iliaca Block as Rescue Analgesia Following Total Hip Arthroplasty
Acronym: SOSBIFSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Principal Investigator, Abderrahmen BARGAOUI, Principal Investigator, Institut Mutualiste Montsouris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANESTH-03-2024; 2024-A02290-47 (Other: ANSM)
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hip Arthroplasty, Total; Post Operative Pain, Acute; Nerve Block
Keywords: Total hip arthroplasty; Regional anesthesia; Nerve blocks; Supra-inguinal fascia iliaca block; Enhanced recovery after surgery; Acute post-operative pain; Rescue analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized, assessor and patient blinded, placebo controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIFIB group (Experimental): The ultrasound probe is placed in a cephalo-caudal orientation, over the inguinal ligament, lateral to the femoral nerve. The iliacus muscle, which is covered caudally by the sartorius muscle and cephalically by the internal oblique muscle, is visualized in depth. Between these two muscles, an area is identified where the iliacus muscle is covered only by subcutaneous tissue. The needle is introduced in a cranio-caudal direction, and the injection is initiated in this area, beneath the fascia iliaca. The needle then advances through the space created by the injection, as far as possible in a cephalic direction, beneath the internal oblique muscle. An injection of 40 ml of 0.1% ropivacaine is administered.
  Interventions: Procedure: Ultrasound guided supra inguinal fascia iliaca block; Procedure: Surgical and anesthetic protocol
- Placebo group (Sham Comparator): Five milliliters of saline are injected subcutaneously under ultrasound guidance
  Interventions: Procedure: Placebo Injection; Procedure: Surgical and anesthetic protocol

INTERVENTIONS:
Procedure: Ultrasound guided supra inguinal fascia iliaca block — The ultrasound probe is placed in a cephalo-caudal orientation, over the inguinal ligament, lateral to the femoral nerve. The iliacus muscle, which is covered caudally by the sartorius muscle and cephalically by the internal oblique muscle, is visualized in depth. Between these two muscles, an area is identified where the iliacus muscle is covered only by subcutaneous tissue. The needle is introduced in a cranio-caudal direction, and the injection is initiated in this area, beneath the fascia iliaca. The needle then advances through the space created by the injection, as far as possible in a cephalic direction, beneath the internal oblique muscle. An injection of 40 ml of 0.1% ropivacaine is administered.
  Arms: SIFIB group
Procedure: Placebo Injection — Five milliliters of saline are injected subcutaneously under ultrasound guidance
  Arms: Placebo group
Procedure: Surgical and anesthetic protocol — All patients receive standard general anesthesia:
  * Induction of anesthesia by sufentanil, ketamine, propofol and tracrium if needed,
  * Maintenance of anesthesia by sevoflurane and sufentanil if needed,
  * Prevention of PONV by dexamethasone and droperidol,
  * Post-operative analgesia by paracetamol, ketoprofene, nefopam, as indicated. Total hip arthroplasty is performed by anterior or postero-lateral approach, depending on surgeon preference.
  In the post-anesthesia care unit, if numerical pain rating scale at rest is >=4, patients are randomized to receive experimental or placebo intervention.

SUMMARY:
Hip replacement surgery is one of the most commonly performed surgical procedures in France, with approximately 150,000 procedures per year. Postoperative recovery has significantly improved in recent years, enabling faster rehabilitation.

Although generally considered moderately painful, hip replacement surgery can, in some difficult-to-predict cases, lead to severe postoperative pain, requiring high doses of morphine, which may cause side effects and delay recovery.

In other surgical procedures, regional anesthesia (nerve blocks) has been successfully used for pain relief. However, its effectiveness after hip replacement surgery has not yet been fully proven.

A recent regional anesthesia technique-the Supra-Inguinal Fascia Iliaca Block (SIFIB)-which numbs a significant portion of the nerves around the hip, has recently been developed.

When performed in all patients undergoing hip arthroplasty, the benefit of this technique could not be demonstrated. In addition, this technique may lead to transcient muscle blockade, wich also can delay recovery.

In order to limit the use of nerve blocks to painful patients, we designed this study where the nerve block is performed only in patients experiencing significant paint after surgery.

In conclusion, this study aims to assess the benefits of performing a rescue SIFIB in the recovery room for patients who experience significant postoperative pain after hip replacement surgery. The evaluation will focus on pain relief and ability to walk.

No new treatment is being tested. The technique uses a commonly administered local anesthetic to numb the nerves.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a primary total hip arthroplasty under general anesthesia,
* written informed consent.

Non inclusion criteria:

* contra indication to ropivacaine
* vulnerable person

Exclusion Criteria:

* per-operative complication making wheight-bearing and walking contra-indicated.
* patient without significant pain post-operatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 2 hours post operatively
  Composite outcome is validated if all of these 3 items are validated:
  * numerical pain rating scale (from 0 to 10) at rest is < 4,
  * and intravenous morphine < 0,1 mg/kg,
  * and first mobilization successful. First mobilization is validated if patient can stand up, walk 5 meters then sit down in a wheelchair.

SECONDARY OUTCOMES:
Morphine consumption | 24 hours post operatively
  oral morphine equivalent needings
Pain evaluation | 6, 12 and 24 hours post operatively
  Numerical pain rating scale (0-10=) at rest Numerical rating scale for pain is described as a scale from a minimum of 0, associated with no pain, to a maximum of 10, associated with the worst possible pain.
Length of hospital stay | An average of 2 to 3 days up to 1 week
  Number of in-hospital post operative nights
Patient satisfaction | Day 1
  Patient satisfaction assessment on pain management, using a 5-degrees Likert scale.
  (1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahmen BARGAOUI, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Zhang XY, Ma JB. The efficacy of fascia iliaca compartment block for pain control after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Jan 25;14(1):33. doi: 10.1186/s13018-018-1053-1. PMID 30683117
- [Background] Changjun C, Xin Z, Yue L, Liyile C, Pengde K. Key Elements of Enhanced Recovery after Total Joint Arthroplasty: A Reanalysis of the Enhanced Recovery after Surgery Guidelines. Orthop Surg. 2023 Mar;15(3):671-678. doi: 10.1111/os.13623. Epub 2023 Jan 3. PMID 36597677
- [Background] Bloc S, Alfonsi P, Belbachir A, Beaussier M, Bouvet L, Campard S, Campion S, Cazenave L, Diemunsch P, Di Maria S, Dufour G, Fabri S, Fletcher D, Garnier M, Godier A, Grillo P, Huet O, Joosten A, Lasocki S, Le Guen M, Le Sache F, Macquer I, Marquis C, de Montblanc J, Maurice-Szamburski A, Nguyen YL, Ruscio L, Zieleskiewicz L, Caillard A, Weiss E. Guidelines on perioperative optimization protocol for the adult patient 2023. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101264. doi: 10.1016/j.accpm.2023.101264. Epub 2023 Jun 7. PMID 37295649
- [Background] Anger M, Valovska T, Beloeil H, Lirk P, Joshi GP, Van de Velde M, Raeder J; PROSPECT Working Group* and the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guideline for total hip arthroplasty: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Aug;76(8):1082-1097. doi: 10.1111/anae.15498. Epub 2021 May 20. PMID 34015859
- [Background] Memtsoudis SG, Cozowicz C, Bekeris J, Bekere D, Liu J, Soffin EM, Mariano ER, Johnson RL, Go G, Hargett MJ, Lee BH, Wendel P, Brouillette M, Kim SJ, Baaklini L, Wetmore DS, Hong G, Goto R, Jivanelli B, Athanassoglou V, Argyra E, Barrington MJ, Borgeat A, De Andres J, El-Boghdadly K, Elkassabany NM, Gautier P, Gerner P, Gonzalez Della Valle A, Goytizolo E, Guo Z, Hogg R, Kehlet H, Kessler P, Kopp S, Lavand'homme P, Macfarlane A, MacLean C, Mantilla C, McIsaac D, McLawhorn A, Neal JM, Parks M, Parvizi J, Peng P, Pichler L, Poeran J, Poultsides L, Schwenk ES, Sites BD, Stundner O, Sun EC, Viscusi E, Votta-Velis EG, Wu CL, YaDeau J, Sharrock NE. Peripheral nerve block anesthesia/analgesia for patients undergoing primary hip and knee arthroplasty: recommendations from the International Consensus on Anesthesia-Related Outcomes after Surgery (ICAROS) group based on a systematic review and meta-analysis of current literature. Reg Anesth Pain Med. 2021 Nov;46(11):971-985. doi: 10.1136/rapm-2021-102750. Epub 2021 Aug 25. PMID 34433647
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233